CLINICAL TRIAL: NCT03425604
Title: Role of Intrauterine Insemination in Patients With Endometriosis I-II
Status: Completed | Type: Observational
Sponsor: IVI Bilbao (Other)
Responsible Party: Sponsor
Other Study IDs: IVIBILBAO
Record Dates: First submitted 2018-02-01; First posted 2018-02-07 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2018-02

CONDITIONS: Endometriosis I-II

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis I y II, according to ASRM classification: Cycles were chosen for analysis only when all the following selection criteria were satisfied: < 38 years old women, antral follicle count > 6, basal FSH < 10mUI/ml, BMI<30, Infertility time <4 years, absence of uterine malformations, endometrial polyps or myomas, absence of known thrombofilia, normal kayotype, < 3 previous IUI cycles, no male severe factor associated
  Interventions: Procedure: Intrauterine insemination
- patients without endometriosis: Cycles were chosen for analysis only when all the following selection criteria were satisfied: < 38 years old women, antral follicle count > 6, basal FSH < 10mUI/ml, BMI<30, Infertility time <4 years, absence of uterine malformations, endometrial polyps or myomas, absence of known thrombofilia, normal kayotype, < 3 previous IUI cycles, no male severe factor associated
  Interventions: Procedure: Intrauterine insemination

INTERVENTIONS:
Procedure: Intrauterine insemination

SUMMARY:
Intrauterine insemination (IUI) is an ART that provides good results in selected patients, improving their reproductive prognosis. Endometriosis I y II, according to ASRM classification, remains an indication to perform IUI. This indication is on continuous debate, considering that different studies have shown controversial results about it, due to the poor reproductive outcomes in this group of patients

ELIGIBILITY:
Inclusion Criteria:< 38 years old women, antral follicle count > 6, basal FSH < 10mUI/ml, BMI<30, Infertility time <4 years, absence of uterine malformations, endometrial polyps or myomas, absence of known thrombofilia, normal kayotype, < 3 previous IUI cycles, no male severe factor associated

-

Exclusion Criteria:

* > 38 years old

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: We analyzed the database (SIVIS) containing information on IUI treatment cycles carried out at the IVI-Clinics between 2011 and 2017.
Sampling Method: Non-Probability Sample
Enrollment: 9979 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
pregnancy rate | 2011-2017
  to compare pregnancy rate between Endometriosis I-II patients (according to ASRM classification) vs. control group (patients without endometriosis) going under an IUI cycle

IPD SHARING:
Plan to Share IPD: No